CLINICAL TRIAL: NCT04863638
Title: A Immunobridging and Immunization Schedules Study of COVID-19 Vaccine (Vero Cell), Inactivated in Population Aged ≥ 60 Years Old and 3-17 Years Old Compared With That in Population Aged 18-59 Years Old
Brief Title: A Immuno-bridging and Immunization Schedules Study of COVID-19 Vaccine (Vero Cell), Inactivated
Acronym: COVID-19
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: China National Biotec Group Company Limited (Industry)
Collaborators: Beijing Institute of Biological Products Co Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: BIBP2020004CN
Record Dates: First submitted 2021-04-27; First posted 2021-04-28 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Covid19
Keywords: SARS-CoV-2; SARS-CoV-2 Vaccine; Coronavirus
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (18):
- A1 aged ≥ 71 (Experimental): 300 subjects age ≥ 71 （A1）receive 3 doses of vaccine
  Interventions: Biological: 3-doses schedule 1 of COVID-19 Vaccine (Vero Cell), Inactivated
- A2 aged ≥ 71 (Experimental): 200 subjects age ≥ 71 （A2）receive 3 doses of vaccine
  Interventions: Biological: 3-doses schedule 2 of COVID-19 Vaccine (Vero Cell), Inactivated
- A3 aged ≥ 71 (Experimental): 200 subjects age ≥ 71 (A3) receive 3 doses of vaccine
  Interventions: Biological: 3-doses schedule 3 of COVID-19 Vaccine (Vero Cell), Inactivated
- B1 aged 60-70 (Experimental): 300 subjects age 60-70 (B1) receive 3 doses of vaccine
  Interventions: Biological: 3-doses schedule 1 of COVID-19 Vaccine (Vero Cell), Inactivated
- B2 aged 60-70 (Experimental): 200 subjects age 60-70 (B2) receive 3 doses of vaccine
  Interventions: Biological: 3-doses schedule 2 of COVID-19 Vaccine (Vero Cell), Inactivated
- B3 aged 60-70 (Experimental): 200 subjects age 60-70 (B3) receive 3 doses of vaccine
  Interventions: Biological: 3-doses schedule 3 of COVID-19 Vaccine (Vero Cell), Inactivated
- C1 aged 18-59 (Experimental): 300 subjects age 18-59 (C1) receive 3 doses of vaccine
  Interventions: Biological: 3-doses schedule 1 of COVID-19 Vaccine (Vero Cell), Inactivated
- C2 aged 18-59 (Experimental): 200 subjects age 18-59 (C2) receive 3 doses of vaccine
  Interventions: Biological: 3-doses schedule 2 of COVID-19 Vaccine (Vero Cell), Inactivated
- C3 aged 18-59 (Experimental): 200 subjects age 18-59 (C3) receive 3 doses of vaccine
  Interventions: Biological: 3-doses schedule 3 of COVID-19 Vaccine (Vero Cell), Inactivated
- C4 aged 18-59 (Experimental): 300 subjects age 18-59 (C4) receive 2 doses of vaccine
  Interventions: Biological: 2 doses of vaccine
- D1 aged 9-17 (Experimental): 300 subjects age 9-17 (D1) receive 3 doses of vaccine
  Interventions: Biological: 3-doses schedule 1 of COVID-19 Vaccine (Vero Cell), Inactivated
- D2 aged 9-17 (Experimental): 200 subjects age 9-17 (D2) receive 3 doses of vaccine
  Interventions: Biological: 3-doses schedule 2 of COVID-19 Vaccine (Vero Cell), Inactivated
- D3 aged 9-17 (Experimental): 200 subjects age 9-17 （D3）receive 3 doses of vaccine
  Interventions: Biological: 3-doses schedule 3 of COVID-19 Vaccine (Vero Cell), Inactivated
- D4 aged 9-17 (Experimental): 300 subjects age 9-17 （D4）receive 2 doses of vaccine
  Interventions: Biological: 2 doses of vaccine
- E1 aged 3-8 (Experimental): 300 subjects age 3-8 （E1） receive 3 doses of vaccine
  Interventions: Biological: 3-doses schedule 1 of COVID-19 Vaccine (Vero Cell), Inactivated
- E2 aged 3-8 (Experimental): 200 subjects age 3-8 （E2）receive 3 doses of vaccine
  Interventions: Biological: 3-doses schedule 2 of COVID-19 Vaccine (Vero Cell), Inactivated
- E3 aged 3-8 (Experimental): 200 subjects age 3-8 （E3）receive 3 doses of vaccine
  Interventions: Biological: 3-doses schedule 3 of COVID-19 Vaccine (Vero Cell), Inactivated
- E4 aged 3-8 (Experimental): 300 subjects age 3-8 （E4）receive 2 doses of vaccine
  Interventions: Biological: 2 doses of vaccine

INTERVENTIONS:
Biological: 3-doses schedule 1 of COVID-19 Vaccine (Vero Cell), Inactivated — the schedule of Day 0, 21, 42
  Arms: A1 aged ≥ 71; B1 aged 60-70; C1 aged 18-59; D1 aged 9-17; E1 aged 3-8
Biological: 3-doses schedule 2 of COVID-19 Vaccine (Vero Cell), Inactivated — the schedule of Day 0, 21, 111
  Arms: A2 aged ≥ 71; B2 aged 60-70; C2 aged 18-59; D2 aged 9-17; E2 aged 3-8
Biological: 3-doses schedule 3 of COVID-19 Vaccine (Vero Cell), Inactivated — the schedule of Day 0, 21, 171
  Arms: A3 aged ≥ 71; B3 aged 60-70; C3 aged 18-59; D3 aged 9-17; E3 aged 3-8
Biological: 2 doses of vaccine — the schedule of Day 0, 21
  Arms: C4 aged 18-59; D4 aged 9-17; E4 aged 3-8

SUMMARY:
This trial is a randomized study to evaluate the immunogenicity of COVID-19 Vaccine (Vero Cell), Inactivated and in population aged 60 years old and 3-17 years old with different schedules compared to that in population aged 18-59 years old with 2-dose schedule. And subjects in the same age are randomly assigned to different immunization schedule groups.

DETAILED DESCRIPTION:
This trial is a randomized study to evaluate the immunogenicity of COVID-19 Vaccine (Vero Cell), Inactivated and in population aged 60 years old and 3-17 years old with different schedules (D0,21,42, D0, 21,111,or D0,21,171)compared to that in population aged 18-59 years old with 2-dose schedule (D0,21). And subjects in the same age are randomly assigned to different immunization schedule groups.

ELIGIBILITY:
Inclusion Criteria:

* Aged 3 years and above (after enrolled, subjects will be allocated according to age).
* By asking for medical history and physical examination, the health condition judged by the investigators is well.
* Female subjects of childbearing age are not nursing or pregnant at the time of enrolment (negative urine pregnancy test) and have no family planning within the first 3 months after enrolment. Effective contraceptive measures have been taken within 2 weeks before inclusion.
* No vaccination history of COVID-19 vaccine before enrollment.
* Be able and willing to complete the whole prescribed study plan.
* With self-ability to understand the study procedures, the informed consent & voluntarily sign an informed consent form and be able to comply with the requirements of the protocol.

Exclusion Criteria:

* Confirmed cases, suspected cases or asymptomatic infections of SAR-CoV-2 infection (check "China Disease Prevention and Control Information System").
* Has a history of SARS, MERS infection (self-report, on-site inquiry).
* >14-year-old subjects axillary temperature ≥37.3℃, ≤14-year-old subjects axillary temperature ≥37.5℃.
* Previous severe allergic reactions to vaccination (such as acute allergic reactions, urticaria, dyspnea, angioneurotic edema or abdominal pain) or allergy to known ingredients of inactivated SARS-CoV-2 vaccine have occurred.
* With severe liver diseases, severe kidney diseases, uncontrollable hypertension (systolic blood pressure ≥160 mmHg, diastolic blood pressure ≥100 mmHg), diabetic complications, malignant tumors, various acute diseases, or acute attack period of chronic diseases.
* Has been diagnosed with congenital or acquired immune deficiency, HIV infection, lymphoma, leukemia or other autoimmune diseases.
* Has a history of convulsion, epilepsy, encephalopathy or mental illness or family history.
* With congenital malformations or developmental disorders, genetic defects, severe malnutrition, etc.
* Has a history of coagulation dysfunction (e.g. Coagulation factor deficiency, coagulation disease).
* Received immunotherapy or inhibitor therapy within 3 months (continuous oral or infusion for more than 14 days).
* Received live attenuated vaccinewithin 1 month before this vaccination, other vaccines are inoculated within 14 days before this vaccination.
* Received blood products within 3 months before enrolment.
* Received other research drugs within 6 months before enrolment.
* Other circumstances judged by investigators are not suitable for this clinical trial.

Min Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 4400 (Actual)
Dates: Start 2021-04-29 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
The Geometric Mean Titer (GMT) of anti-SARS-CoV-2 neutralizing antibody | 14 days after the full course immunization
  Neutralizing antibody assay will be performed using the Microcytopathic assay
The four-fold increase rate of anti-SARS-CoV-2 neutralizing antibody | 14 days after the full course immunization
  ≥4 fold increase from baseline

SECONDARY OUTCOMES:
The Geometric Mean Titer (GMT) of anti-SARS-CoV-2 neutralizing antibody | 14 days after the second dose in schedule of Day 0,21,42
  Neutralizing antibody assay will be performed using the Microcytopathic assay
The four-fold increase rate of anti-SARS-CoV-2 neutralizing antibody | 14 days after the second dose in schedule of Day 0,21,42
  ≥4 fold increase from baseline
The Geometric Mean Titer (GMT) of anti-SARS-CoV-2 neutralizing antibody | before the third dose in schedules of Day 0,21,111 and Day 0,21,171
  Neutralizing antibody assay will be performed using the Microcytopathic assay
The four-fold increase rate of anti-SARS-CoV-2 neutralizing antibody | before the third dose in schedules of Day 0,21,111 and Day 0,21,171
  ≥4 fold increase from baseline
Immune Persistence | 3 months, 6 months, 12 months after the full course immunization
  Neutralizing antibody assay will be performed using the Microcytopathic assay
Safety index-Incidence of adverse reactions | From the beginning of the vaccination to 28 days after the full course immunization
  collect the all the adverse events using dairy card and contact card
Safety index-Incidence of serious adverse events | From the beginning of the vaccination to 6 months after the full course immunization
  All SAEs will be collected

OTHER OUTCOMES:
Immune Persistence | 18 months and 24 months after the full immunization
  Neutralizing antibody assay will be performed using the Microcytopathic assay

CONTACTS AND LOCATIONS:
Overall Officials: Yanxia Wang, Bachelor, Principal Investigator — Henan Provincial Center for Disease Control and Prevention
Locations (1):
- Yanjin County Center for Disease Control and Prevention, Xinxiang, Henan, China